CLINICAL TRIAL: NCT02669901
Title: Naloxone Auto-injector as a Universal Precaution for Patients With Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Kaleo Inc. (Other)
Responsible Party: Principal Investigator, Joanna G Katzman, Dr. Joanna Katzman, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-616
Record Dates: First submitted 2015-12-21; First posted 2016-02-01 (Estimated); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Opiate Antagonist Overdose; Opioid-Related Disorders
Keywords: Opioid-Related Disorders; Naloxone; Harm Reduction; Drug Overdose Deaths; Opioid Misuse; Naloxone Coprescribing; Universal Precautions; Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with opioid use disorder (Other): All participants received Naloxone autoinjector as a preventative tool for accidental opioid overdose
  Interventions: Behavioral: Naloxone Auto-Injector

INTERVENTIONS:
Behavioral: Naloxone Auto-Injector — Naloxone auto-injector is FDA approved and labeled for use by family members or caregivers for emergency therapy and rescue wherever opioids are present. Bystanders of patient are able to provide naloxone when drug overdose occurs.

SUMMARY:
The purpose of this pilot-study is to to distribute naloxone auto-injector in a "Universal Precaution" manner to patients with opioid substance use disorder. The objectives are to decrease the number of fatal and nonfatal overdose deaths, to examine and understand the risk factors for serious opioid toxicity and overdose, and to evaluate the unintentional opioid overdose risk utilizing an evidence-based screening questionnaire.

DETAILED DESCRIPTION:
Between April 4, 2016, and May 16, 2017, 395 study participants voluntarily enrolled at the UNM ASAP for this prospective cohort study. The study closed 1 year after enrollment, on May 17, 2018. These study participants were current patients of the University of New Mexico's Addiction and Substance Abuse Program.

This study was approved by the University of New Mexico Human Research and Review Committee and was registered in the National Institutes of Health Clinical Trials (ClinicalTrials.gov Identifier NCT02669901). A certificate of confidentiality is on record at the National Institutes of Health for this study. Written informed consent was obtained from each individual study participant. This study follows the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) reporting guideline.

Each study participant completed the initial visit and at least 1 follow-up visit. Inclusion criteria included history of OUD treated with methadone, buprenorphine, or naltrexone and age 18 years or older. Exclusion criteria included allergy to naloxone and age younger than 18 years.

The UNM ASAP is a federally qualified opioid treatment program (OTP) that provides medication-assisted treatment and behavioral therapy for adults, including pregnant women, as well as adolescents. Approximately 65% of the UNM ASAP patients are women. Most (80%) of the patients had previously used heroin (compared with prescription opioids) as their drug of choice before beginning medication-assisted treatment.

Initial Visit Data Collection At the initial visit, study participants provided demographic data, social history, limited medical history, type of medication-assisted treatment, medication list, and history of illicit drug use.21 All 395 study participants enrolled were evaluated to determine whether they had received a naloxone prescription in the year before enrollment. First, each participant's electronic medical record was queried to see whether a prescription for naloxone was written in the year before study enrollment. Second, every study participant was personally asked by the research coordinator at the initial study visit whether they had directly received a naloxone prescription in the year before enrollment.

OD Education and Naloxone Distribution During the initial visit, the study participant along with his or her companion, if present, were provided with OD information and learned the importance of using naloxone. Study participants were encouraged, but not required, to bring a companion to the visit. The education included recognizing signs and symptoms of an OD, the importance of calling 911, rescue breathing techniques, and staying with the person experiencing the OD until medical help has arrived. The research coordinator distributed 1 naloxone kit (2 doses) to study participants after they felt confident with using the naloxone autoinjector.21,22 Study participants were informed that they could return to the clinic to obtain a naloxone replacement kit if needed.

Quarterly Follow-up Visits Every 3 months, study participants were asked to follow up with the study coordinator to report on whether an OD reversal was performed and whether naloxone replacement kits were needed. Study participants could also obtain naloxone replacement kits Monday through Friday during clinic hours (7 am to 5 pm). Urine toxicology screens were obtained as part of the routine UNM ASAP clinic procedure and were reported previously.23

Statistical Analysis Stata statistical software version 15 (Stata Corp) was used for all analyses, including distributions of study participants' characteristics at the initial visit, relationships between community members for whom OD reversal was performed and study participants, number of OD reversals performed, and reasons for replacement of THN kits. Stata 15 was also used for χ2 tests for statistical significance of associations between companion attendance at initial opioid education and performing at least 1 OD reversal. One-sided P < .05 was considered statistically significant. Data analysis was performed from May 2018 to July 2019.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with methadone, naltrexone or buprenorphine as medication assisted treatment at the UNM Addiction and Substance Abuse Program (UNM ASAP) aged 18 or older

Exclusion Criteria:

* Subjects who are allergic to naloxone and its inactive ingredients. Inactive ingredients include buffering agents.
* Subjects younger than 18.
* Subjects not being treated at UNM ASAP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Katzman, MD, Principal Investigator — University of New Mexico School of Medicine
Locations (1):
- UNM Hospitals - Alcohol and Substance Abuse Program, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
We published our study results. Please refer to the following publications:
  PMID: 32101312 PMID: 32404109 PMID: 29227321 PMID: 32600618 PMID: 30303890

REFERENCES:
- [Background] Katzman JG, Takeda MY, Greenberg N, Moya Balasch M, Alchbli A, Katzman WG, Salvador JG, Bhatt SR. Association of Take-Home Naloxone and Opioid Overdose Reversals Performed by Patients in an Opioid Treatment Program. JAMA Netw Open. 2020 Feb 5;3(2):e200117. doi: 10.1001/jamanetworkopen.2020.0117. PMID 32101312

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Opioid Substance Abuse Disorders: All participants received Naloxone autoinjector as a preventative tool for accidental opioid overdose.
Period: Overall Study
Arm/Group | Patients With Opioid Substance Abuse Disorders
Started | 395
Completed | 336
Not Completed | 59

BASELINE CHARACTERISTICS:
Groups:
- Patients With Opioid Substance Abuse Disorders: The study participants received 2 (two) 0.4 mg of naloxone auto-injectors (intramuscular injection). The participants were instructed to use the naloxone autoinjector when they witnessed an opioid overdose. Also, they were instructed to educate their bystanders on what opioid overdose is and asked them to use naloxone in case of their opioid overdose. The auto-injectors could be used twice if one injection was not sufficient for an opioid overdose.
Arm/Group | Patients With Opioid Substance Abuse Disorders
Number analyzed (Participants) | 395
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 270
  Male | 125
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 16
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 360
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 395
Medication-assisted treatment [Count of Participants; unit: Participants]
  Methadone | 279
  Buprenorphine | 109
  Naltrexone (oral or intramuscular) | 7
Companion for naloxone education [Count of Participants; unit: Participants]
  Present | 33
  Not present | 354
  Unknown | 8

OUTCOME MEASURES:

1. Primary Outcome: To Measure the Association of Take-home Naloxone With Overdose Reversals Performed by Patients With Opioid Use Disorder Enrolled in an Opioid Treatment Program
Description: The study participants received 2 naloxone kits at their initial visit. They were educated on how to recognize the signs and symptoms of an OD, the importance of calling 911, rescue breathing techniques, and staying with the person experiencing the OD until medical help has arrived. They were asked about their use of naloxone every 3 months, including the situation of the naloxone kits, dose, and to whom they used.
Time Frame: 1 year after enrollment
Population: Study participants who completed at least 1 follow up visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Opioid Use Disorder
Number analyzed (Participants) | 336
Participants
  Study participants who reported OD reversa | 73
  Study participants who reported no OD reversals | 263

ADVERSE EVENTS:
Time Frame: 1 year after enrollment
Description: Because the naloxone kits were used to rescue community people with OD, no adverse events were reported in the patients among the study participants who received the naloxone kits. Because adverse events were self-reported, the investigators had limitations in verifying the information from the study participants.
Groups:
- Patients With Opioid Use Disorder: The study participants reported that they did not observe adverse events when using the naloxone auto-injectors for people with opioid overdose.
Arm/Group | Patients With Opioid Use Disorder
All-Cause Mortality (participants affected / at risk) | 0/395
Serious Adverse Events (participants affected / at risk) | 0/395
Other Adverse Events (participants affected / at risk) | 0/395

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT02669901/Prot_SAP_000.pdf